CLINICAL TRIAL: NCT01387438
Title: Cross-sectional Study on the Incidence,Factors,and Importance of Brown Adipose Tissue in Adult Chinese
Brief Title: The Incidence,Factors,and Importance of Brown Adipose Tissue in Chinese Adults
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Yiming Li, Huashan Hospital
Other Study IDs: KY2009-279
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2009-11

CONDITIONS: Obesity
Keywords: Brown Adipose Tissue; Cross sectional study; Chinese Adults; Factor
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Previous studies have shown that active brown adipose tissue (BAT) is present in adults and may play important roles in material and energy metabolism. However, most of these studies were tumor-based populations and retrospective study. Due to the large amount in our cohort, the investigators are able to promote a cross-sectional study of the incidence and factors of BAT in adult chinese. In addition, the investigators can analyse the metabolic profiles in healthy adults with active BAT.

DETAILED DESCRIPTION:
The investigators will perform a cross sectional analysis on the chinese adults who use 18F-fluorodeoxyglucose positron emission tomography/computed tomography (PET/CT) to scan the whole body at Huashan Hospital from 2009 to 2013. BAT activity will be measured by PET/CT. Not only demographic data on sex, age, medication and medical history,but also data on body composition and physical examination will be collected for all subjects. Imaging date,outdoor temperature and fasting blood samples will be collected as well. In addition, the investigators will analyse the metabolic profiles in healthy adults with active BAT and their negative controls,such as lipid profiles,fasting glucose and insulin sensitivity, adipokines and other biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with detectable brown adipose tissue
* Negative controls,consisting of one subject who underwent PET/CT scans at the same day but without detectable BAT

Exclusion Criteria:

* Younger than 18 years
* Pregnant women
* With implantable medical electronic instrument

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent scanning PET-CT at Huashan Hospital Medical Centre from 2009 to 2013
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, Doctor, Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China